CLINICAL TRIAL: NCT06859814
Title: Value of Infection Control Programs on Infection Associated with Urinary Tract Catheterization in Sohag University Hospital
Acronym: Urinary tract
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Mosleh, Mohamed mahmoud mohamed, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Soh-Med--25-2-01MS
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: UTI
Keywords: UTI; Urinary catheterization
MeSH Terms: interventions — Urinary Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with urinary catheters (Experimental): Adult patients (≥ 18 years) who are catheterized during their hospitalization.
  Interventions: Procedure: urinary catheterization

INTERVENTIONS:
Procedure: urinary catheterization — urine samples for culture and sensitivity will be collected in patients having urinary tract infection and we will use sterile container 50cc for urine sampling culture on blood or macconkey medium for detection type of organism .

SUMMARY:
The aim of this study is to evaluate the effectiveness of an infection control program implemented at Sohag University Hospital in reducing the incidence of catheter-associated urinary tract infections (CAUTIs) among patients requiring urinary catheterization.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (≥ 18 years) who are catheterized during their hospitalization. Patients who provide informed consent to participate in the study.

Exclusion Criteria:

Patients with a known history of urinary tract infections prior to hospitalization.

Patients who have indwelling catheters for more than 14 days before the study. Patients with urinary tract anomalies or other conditions that may affect infection rates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of CAUTIs: | one month
  The primary outcome will be the rate of CAUTIs before and after the implementation of the infection control program. CAUTIs will be defined according to the criteria established by the Centers for Disease Control and Prevention (CDC) and will include clinical signs, symptoms, and positive urine cultures.

SECONDARY OUTCOMES:
Length of Hospital Stay: | one month
  The average length of stay for patients with CAUTIs will be compared preand post-intervention. A reduction in length of stay may indicate improved patient outcomes and decreased complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospitals, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided